CLINICAL TRIAL: NCT05524857
Title: Phase I Trial of Fedratinib in Combination With Decitabine in Patients With Myeloproliferative Neoplasms in Accelerated and Blast Phase
Brief Title: Combination of Fedratinib and Decitabine for Myeloproliferative Neoplasms (MPN)- Accelerated Phase (AP)/Blast Phase (BP)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Closed by Sponsor
Sponsor: Joseph Jurcic (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor-Investigator, Joseph Jurcic, Professor of Medicine, Columbia University
Organization: Columbia University (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AAAT9407
Record Dates: First submitted 2022-08-30; First posted 2022-09-01 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Myeloproliferative Neoplasm
Keywords: Blast Phase; Fedratinib; Decitabine
MeSH Terms: conditions — Myeloproliferative Disorders; Blast Crisis | interventions — fedratinib; Decitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fedratinib 300 mg (Experimental): Cohort 1: 300 mg of Fedratinib by mouth, once daily during each 28-day cycle
  Interventions: Drug: Fedratinib Oral Capsule 300 mg; Drug: Decitabine 20 mg/m2
- Fedratinib 400 mg (Experimental): Cohort 2: 400 mg of Fedratinib by mouth, once daily during each 28-day cycle
  Interventions: Drug: Decitabine 20 mg/m2; Drug: Fedratinib Oral Capsule 400 mg

INTERVENTIONS:
Drug: Fedratinib Oral Capsule 300 mg — 300 mg by mouth, once daily
  Other Names: Inrebic
  Arms: Fedratinib 300 mg
Drug: Decitabine 20 mg/m2 — 20 mg/m2 for injection, for intravenous use
  Other Names: Dacogen
Drug: Fedratinib Oral Capsule 400 mg — 400 mg by mouth, once daily
  Other Names: Inrebic
  Arms: Fedratinib 400 mg

SUMMARY:
The purpose of this research is to study the safety and tolerability and to establish the maximum tolerated dose (MTD) of the combination of two drugs, fedratinib and decitabine, for the treatment of advanced-phase MPNs.

DETAILED DESCRIPTION:
This is a single center phase I dose-escalation trial of Fedratinib in Combination with Decitabine in Patients with Myeloproliferative Neoplasms. The primary objective is to determine the maximum tolerated dose of the combination therapy, using a 3+3 dose escalation algorithm. Fedratinib will be administered at 2 dose levels: 300 mg and 400 mg by mouth, once daily. Fedratinib will be administered concomitantly with decitabine 20 mg/m2 intravenously over 1 hour per day for 5 days in 28-day cycles.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have MPN-AP as defined by 10%-19% blasts in the peripheral blood or bone marrow and evidence of dysplastic marrow features with a concomitant diagnosis of essential thrombocythemia (ET), polycythemia vera (PV) or primary myelofibrosis (PMF) or a diagnosis of MPN-BP as defined by 20% blasts in the blood or bone marrow following a previous diagnosis of ET, PV or PMF.
* Subjects must have adequate organ function documented within 14 days of study entry as follows:

  1. Estimated creatinine clearance (by Cockcroft-Gault Equation) of ≥ 50 mL/min
  2. Serum total bilirubin ≤ 1.5 × ULN (unless attributable to Gilbert's disease or hemolysis, in which case the direct bilirubin level must be ≤ 1.5 × upper limit of normal (ULN)).
  3. Alkaline phosphatase, serum aspartate aminotransferase (AST) and alanine transaminase (ALT) ≤ 2.5 × ULN.
* ≥ 18 years of age.
* Eastern Cooperative Oncology Group (ECOG) Performance status of 0-2. Patients with ECOG performance status of 3 will be eligible if the lower performance status is deemed by the investigator to be due entirely to MPN-AP/BP and not due to another comorbidity.

Exclusion Criteria:

* Receipt of chemotherapy or investigational therapy, with the exception of hydroxyurea, within 4 weeks of study entry. Previous treatment at any time with decitabine, fedratinib or ruxolitinib as single agents will not exclude eligibility. Previous stem cell transplant will not exclude eligibility as long as other inclusion/exclusion criteria have been met and subjects do not have Grade ≥ II graft-versus-host disease (GVHD) requiring systemic immunosuppressive therapy.
* Subjects with an Human leukocyte antigen (HLA)-compatible donor or stem cell source who are immediate candidates for allogeneic hematopoietic cell transplantation (HCT).
* Subjects who are receiving any concurrent treatment for acute myeloid leukemia (AML), including other investigational agents.
* Diagnosis of acute myelofibrosis.
* Uncontrolled intercurrent illness including, but not limited to hepatitis, human immunodeficiency virus (HIV)-positive subjects receiving combination antiretroviral therapy, ongoing or active infection, symptomatic congestive heart failure (New York Heart Association Class 3 or 4), unstable angina pectoris, ventricular arrhythmia, Child-Pugh Class C cirrhosis, or psychiatric illness/social situations that would limit compliance with study requirements.
* Subjects with a prior history of Wernicke's encephalopathy (WE) will be excluded. If a subject has signs or symptoms of encephalopathy, including Wernicke's encephalopathy (e.g. severe ataxia, ocular paralysis or cerebellar signs), thiamine deficiency must be excluded and a brain MRI should be obtained prior to study initiation to evaluate for WE.
* Other medications, severe acute/chronic medical or psychiatric conditions, or laboratory abnormalities that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results, that in the judgment of the Investigator would make the subject inappropriate for entry into this study.
* Pregnant women are excluded because of the potential for teratogenic or abortifacient effects.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2022-01-28 (Actual); Primary Completion 2024-04-09 (Actual); Study Completion 2024-04-09 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of Decitabine and Fedratinib | Up to 8 weeks for each dosing cohort
  The MTD will be determined using a 3+3 algorithm. If < 33% of the subjects enrolled at a dose level experience a dose-limiting toxicity (DLT), escalation to the next designated dose cohort will continue. If ≥ 33% of the subjects enrolled at a dose level experience a DLT, the previous dosing cohort will be considered the MTD. DLT is defined as: (1) Grade 3, 4, or 5 non-hematologic toxicity considered at least possibly related to the study drug, except for infection, bleeding, fever, fatigue, dyspnea, and (2) Grade 3, 4, or 5 anemia, neutropenia or thrombocytopenia with a hypocellular bone marrow and < 5% marrow blasts lasting for 42 days or more.

SECONDARY OUTCOMES:
Complete Remission (CR) Rate | Up to 3 years
  Complete remission defined as participants that are free of all symptoms related to leukemia and have an absolute neutrophil count ≥ 1 x 10^9/L, no need for red blood cell transfusion, platelet count ≥ 100 x 10^9/L, and normal marrow differential (≤ 5 % blasts) in a normo- or hypercellular marrow.
Composite Complete Remission (CRc) Rate | Up to 3 years
  CRc defined as (CR + Complete remission with incomplete count recovery (CRi)). CRi defined as CR but incomplete count recovery (absolute neutrophil count < 1000/microL or platelet count < 100,000/micro/L).
Partial Remission (PR) Rate | Up to 3 years
  PR defined as CR with 6 - 25 % abnormal cells in the marrow or 50 % decrease in bone marrow blasts.
Progression Free Survival (PFS) | Up to 3 years
  PFS is defined as the duration of time from entry on study to time of recurrence, flow cytometric relapse, cytogenetic relapse, molecular relapse, or death, whichever occurs first.
Overall Survival (OS) | Up to 3 years
  OS is defined as the duration of time from entry on study to time of death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Jurcic, MD, Principal Investigator — Columbia University
Locations (1):
- New York Presbyterian Hospital/Columbia University Irving Medical Center, New York, New York, United States